CLINICAL TRIAL: NCT05394870
Title: Clinical and Electrophysiological Evaluation of the Effectiveness of Manual Lymphatic Drainage in Patients With Mild-to-moderate Carpal Tunnel Syndrome
Brief Title: Clinical and Electrophysiological Evaluation of the Effectiveness for Manual Lymphatic Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Lecturer, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-03.02
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Carpal Tunnel Syndrome; Electrophysical Evaluation; Manual Lymphatic Drainage
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Manual Lymphatic Drainage; Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: manual lymphatic drainage (massage); Other: Splint treatment
- control group (Active Comparator)
  Interventions: Other: Splint treatment

INTERVENTIONS:
Other: manual lymphatic drainage (massage) — Patients will begin treatment with manual lymphatic drainage in the affected extremity. In this context, while the patients are in the supine hook position, lymph drainage will be applied first to the neck and then to the abdomen. After the stimulation of the central lymph nodes, the lymph circulation will be increased by stimulating the axillary lymph nodes of the relevant region. First, the proximal part will be drained and it will be advanced towards the distal. Drainage will be repeated depending on the edema at the distal forearm-wrist level.
  Arms: study group
Other: Splint treatment — The splint routinely given to patients diagnosed with mild to moderate carpal tunnel syndrome will be given to both groups in these patients

SUMMARY:
When the other usage areas of the manual lymphatic drainage technique in the literature, except for the treatment of lymphedema, were examined recently, it was seen that it was also applied in orthopedic and neurological cases in a limited number of studies. The aim of our study is to investigate the effectiveness of manual lymphatic drainage on clinical and electrophysiological findings in carpal tunnel syndrome

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate carpal tunnel syndrome on electrodiagnostic examination
* Being between 20-55 years old
* Volunteering to participate in the treatment to be given

Exclusion Criteria:

* Have a systemic inflammatory disease
* Having any disease that may cause polyneuropathy, such as diabetes mellitus
* Cognitive impairment
* Receiving psychotherapy
* Having a pacemaker
* illiterate
* Having a disease affecting the central nervous system
* Having a hearing problem
* Any skin disease that would contraindicate manual lymphatic drainage
* Arterial or venous circulation disorder that would contraindicate manual lymphatic drainage

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold | 15 minutes
  Each evaluation will be repeated 3 times with 10 seconds between measurements, and the data will be recorded by taking the average of the last two measurements (15). The patients will be evaluated by measuring the transverse carpal ligament, radioulnar joint and extensor digitorum muscle with an algometer before and at the end of the treatment. measurements will be recorded in kg/cm2
Boston Carpal Tunnel Questionnaire (BCTQ) | 10 minutes
  BCTQ, a self-report measure of CTS, evaluates two domains: 1. The symptom severity scale (BCTQSS) has 11 items that assess pain, paresthesia, and weakness. 2. The functional status scale (BCTQ-FS) evaluates the ability to perform manual activities with 8 items. Each item evaluates the increasing severity of symptoms or difficulty with a high score.
Electrodiagnostic evaluation | 15 minutes
  Median motor nerve latency, median motor nerve conduction velocity, compound muscle action potential amplitude will be measured at both levels. Median sensory nerve conduction studies will be performed by antidromic recording with a superficial electrode from the 3rd finger and a stimulus will be given from the wrist 14 cm proximal. Median sensory nerve latency, median sensory nerve conduction velocity and sensory nerve action potential will be calculated for both applications. nerve potentials will be calculated in m/sec

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Science University, Kütahya, Centrum, Turkey (Türkiye)

REFERENCES:
- [Derived] Akdeniz Leblebicier M, Cihan E, Yaman F, Sahbaz Pirincci C, Ture A, Kavuncu V. Can manual lymphatic drainage be a new treatment option in mild-moderate carpal tunnel syndrome? A randomized controlled study. J Hand Ther. 2025 Jul-Sep;38(3):584-593. doi: 10.1016/j.jht.2024.12.020. Epub 2025 Feb 6. PMID 39919926